CLINICAL TRIAL: NCT04073342
Title: Inflammatory Mediators and Intestinal Genes Expression Associated With Necrotizing Enterocolitis in Preterm Infants
Brief Title: Intestinal Genes Expression Associated With Necrotizing Enterocolitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ASAli, Assistant lecturer of pediatric and neonatology , principle investigator,clinical doctor, Assiut University
Other Study IDs: gene expression in necrotizing
Record Dates: First submitted 2019-08-27; First posted 2019-08-29 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-08

CONDITIONS: Neonatal Disease
MeSH Terms: conditions — Infant, Newborn, Diseases | interventions — Interleukin-8

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgical Necrotizing enterocolitis: Cases of preterm infants with necrotizing enterocolitis need surgical intervention
  Interventions: Genetic: Gene expression of inflammatory mediator (Interleukin 8) and recognition receptor of Toll like receptor (TLR4).
- Non Necrotizing enterocolitis: babies with intestinal operations for non necrotizing enterocolitis pathologies like congenital intestinal obstruction.
  Interventions: Genetic: Gene expression of inflammatory mediator (Interleukin 8) and recognition receptor of Toll like receptor (TLR4).

INTERVENTIONS:
Genetic: Gene expression of inflammatory mediator (Interleukin 8) and recognition receptor of Toll like receptor (TLR4). — Ileal tissue from both group will be tested for gene expression of inflammatory mediator (Interleukin 8) and recognition receptor of Toll like receptor (TLR4).

SUMMARY:
In recent days, necrotizing enterocolitis is one of the most common and devastating problem in preterm infants. Therefore, it became a high growing research topic in the last decade.

The development of medical care increases the survival of preterm babies and consequently increase the number of cases with this serious problem. A systematic review shows the incidence of necrotizing enterocolitis is about 2-7% in babies less than 32weeks gestation and 5-22% in baby's birth weight less than 1000gram.

DETAILED DESCRIPTION:
In 2011, study on average cost of necrotizing enterocolitis in United States shows average cost of health service for preterm baby without necrotizing enterocolitis and with necrotizing enterocolitis 74,004 $-198,040 $ respectively.Babies surviving from necrotizing enterocolitis are at risk of long term complication such as short bowel syndrome and intestinal stricture.Furthermore, impairment of neurodevelopment and growth are usually observed in these babies.In spite of decades of researches on the disease, pathogenesis of necrotizing enterocolitis still unclear. We still don't know how to prevent and treat the disease. However, advancement of researches in the field of microbiology and cellular biology of the intestine of preterm infants could lead to more understanding for early diagnosis, prevention and proper treatment. Enteral feeding in preterm pigs lead to upregulation of inflammatory and pattern recognition receptor genes including interleukin8 and Toll like receptor-4 with corresponding condensation of chromatin configuration that lead to initiation of inflammatory process and development of necrotizing enterocolitis. It is not known if these changes are present in human preterm bowel.T cell effector function in preterm infant immune response is characterised by preponderance of interleukin-8 producing T-cells and has the potential to activate neutrophils and γδ T cells.γδ T cells are predominant intra-epithelial lymphocyte in immature preterm gut and has a role in maintaining intestinal integrity.

ELIGIBILITY:
Inclusion Criteria:

* Cases of necrotizing enterocolitis diagnosed by modified Bells criteria, radiological picture and need surgical intervention.

Exclusion Criteria:

* Cases of severe intrauterine growth retardation.
* Cases with severe congenital anomalies.

Ages: 1 Day to 30 Days | Sex: All
Age Groups: Child
Study Population: Surgical cases of necrotizing enterocolitis and control from babies with intestinal operations for non necrotizing enterocolitis pathology (preterm and term infants).
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Intestinal gene expression | 2 years
  Intestinal gene expression of interleukin 8
Toll like receptor 4 | 2 years
  Gene expression of Toll like receptor 4 in cases of necrotizing enterocolitis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Battersby C, Santhalingam T, Costeloe K, Modi N. Incidence of neonatal necrotising enterocolitis in high-income countries: a systematic review. Arch Dis Child Fetal Neonatal Ed. 2018 Mar;103(2):F182-F189. doi: 10.1136/archdischild-2017-313880. Epub 2018 Jan 9. PMID 29317459
- [Background] Ganapathy V, Hay JW, Kim JH. Costs of necrotizing enterocolitis and cost-effectiveness of exclusively human milk-based products in feeding extremely premature infants. Breastfeed Med. 2012 Feb;7(1):29-37. doi: 10.1089/bfm.2011.0002. Epub 2011 Jun 30. PMID 21718117
- [Background] Federici S, De Biagi L. Long Term Outcome of Infants with NEC. Curr Pediatr Rev. 2019;15(2):111-114. doi: 10.2174/1573396315666181130144925. PMID 30499415
- [Background] Willems R, Krych L, Rybicki V, Jiang P, Sangild PT, Shen RL, Hensel KO, Wirth S, Postberg J, Jenke AC. Introducing enteral feeding induces intestinal subclinical inflammation and respective chromatin changes in preterm pigs. Epigenomics. 2015;7(4):553-65. doi: 10.2217/epi.15.13. PMID 26111029
- [Background] Gibbons D, Fleming P, Virasami A, Michel ML, Sebire NJ, Costeloe K, Carr R, Klein N, Hayday A. Interleukin-8 (CXCL8) production is a signatory T cell effector function of human newborn infants. Nat Med. 2014 Oct;20(10):1206-10. doi: 10.1038/nm.3670. Epub 2014 Sep 21. PMID 25242415